CLINICAL TRIAL: NCT00405405
Title: A Phase I Study of the Combination of Chemoradiotherapy With Biologic Therapy for Advanced Head and Neck Cancer
Brief Title: Phase I of Biologics and Chemoradiation Therapy for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06C.46; 2005-58 (Other: CCRRC); 06C.46 (Other: JeffTrial Number)
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Head and Neck Cancer; Parotid Gland Cancer; Thyroid Gland Cancer; Melanoma; Stage IV Head and Neck Cancer
Keywords: Head and neck cancer; Parotid gland cancer; thyroid gland cancer; melanoma; Chemoradiotherapy; bevacizumab; erlotinib
MeSH Terms: conditions — Head and Neck Neoplasms; Parotid Neoplasms; Thyroid Neoplasms; Melanoma | interventions — Cisplatin; Docetaxel; Bevacizumab; Erlotinib Hydrochloride; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): A combination of Cisplatin, Docetaxel, Bevacizumab, Erlotinib, and Radiotherapy
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Drug: Bevacizumab; Drug: Erlotinib; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Cisplatin — * Two cycles during neoadjuvant therapy
  * Response assessment at approximately day 36
  * Concurrent biochemoradiotherapy
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II); CDDP; Platinol; Platinol-AQ
Drug: Docetaxel — * Two cycles during neoadjuvant therapy
  * Response assessment at approximately day 36
  * Concurrent biochemoradiotherapy
  Other Names: Taxotere
Drug: Bevacizumab — * Two cycles during neoadjuvant therapy
  * Response assessment at approximately day 36
  * Concurrent biochemoradiotherapy
  Other Names: Avastin
Drug: Erlotinib — * Two cycles during neoadjuvant therapy (dose escalation)
  * Response assessment at approximately day 36
  * Concurrent biochemoradiotherapy
  Other Names: Erlotinib hydrochloride; Tarceva
Radiation: Radiotherapy — Radiotherapy begins as soon as possible following neoadjuvant chemotherapy, and continues for 7 weeks
  Other Names: Radiation therapy; Radiation oncology; XRT

SUMMARY:
To determine a safe and effective doses of two biologic drugs, erlotinib and bevacizumab when used with chemotherapy and radiation therapy in advanced head and neck cancer

DETAILED DESCRIPTION:
Locally advanced non-operative, Stage IV head and neck cancer has at best a guarded prognosis. Improvements in outcome have been achieved via the combination of chemotherapy and radiotherapy. Concurrent chemoradiotherapy is needed to optimize results, although recent data suggest a benefit from induction therapy as well. Nonetheless, despite high remission rates, most of these patients will suffer local-regional and/or distant recurrence from their disease.

The proposed study will build upon the framework of chemoradiotherapy (induction plus concurrent) via the addition of a double biologic therapy. Specifically, the combination of bevacizumab and erlotinib will be used, as has been studied in other types of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced Carcinoma (epithelial malignancy) of the head and neck. This may include non-squamous carcinomas (e.g. parotid, thyroid, melanoma) in which a large portion of mucosa of the oral cavity and/or laryngopharynx is expected to be irradiated.
* Stage IV disease (T4Nany or TanyN2-3).
* "Oligometastatic" disease is allowable if it is asymptomatic.
* Measurable disease is not required; patients who have had surgical resection are eligible provided that it is felt that the likelihood of cure with conventional postoperative therapy is <40% and provided that there will be at least 28 days from the date of surgery to the start of study therapy.
* Performance status 0-1.
* Creatinine < or = 1.5 mg/dl.
* ANC > or = 1,800 cells/mm3.
* Platelets > or = 150,000 cells/mm3.
* Hemoglobin > or = 10 g/dl (transfusion is acceptable if needed).
* SGOT and/or SGPT < or = 2.5 times the upper institutional limit of normal.
* INR < or = 2.0.
* Age > or = 18 (informed consent).

Exclusion Criteria:

* Current, recent (within 4 weeks of the Day 1, the first infusion of drug in this study) or planned participation in an experimental drug study other than this one.
* Poorly controlled blood pressure, defined as systolic bp > 150 and/or diastolic bp > 100 despite medication.
* Unstable angina.
* NY Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or stroke within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Presence of brain or spinal cord metastases.
* Major surgical procedure(s), open biopsy or significant traumatic injury within 28 days prior to Day 1 (1st day of study treatment) and/or anticipation of need for major surgical procedure during the course of the study.
* Urine protein: Creatinine ratio > or = 1.0 at screening.*
* Carotid artery exposure or other signs of impending carotid artery hemorrhage.
* History of abdominal fistula and/or gastrointestinal abdominal abscess within 6 months prior to enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Prior irradiation that would result in radiotherapy field "overlap."
* Requirement for high dose oral anticoagulation (i.e., goal INR > 2.0). "Mini-dose" anticoagulation as may be used to assist in patency of central venous lines is acceptable. Subcutaneous Low-molecular weight heparin is allowable.
* No known allergies to any of the drug therapies being used in this protocol.
* No pregnancy, lactation or inability to use medically acceptable birth control if of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Bevacizumab and Erlotinib Combined with Chemoradiotherapy for the Treatment of Advanced Head and Neck Cancer | Day 36
  To determine if bevacizumab and erlotinib can be safely combined with chemoradiotherapy for advanced head and neck cancer.

SECONDARY OUTCOMES:
Determination of Dose Limiting Toxicity (DTL) | 30 days
  To determine the appropriate dosing strategy for bevacizumab/erlotinib when combined with chemoradiotherapy for advanced head and neck cancer.
Complete Remission Rate | 6 months
  To obtain preliminary data on the complete remission rate for this treatment combination.

CONTACTS AND LOCATIONS:
Overall Officials: Pramila Rani Anne, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org